CLINICAL TRIAL: NCT00705562
Title: Tolerance of Healthy Term Infants Fed Infant Formulas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK62
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Infant, Newborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Experimental milk protein based infant formula with varying carbohydrate and protein source
  Interventions: Other: milk protein formulas, varying carbohydrate/protein sources
- 2 (Experimental): Experimental milk protein based infant formula with varying carbohydrate and protein source
  Interventions: Other: milk protein formulas, varying carbohydrate/protein sources
- 3 (Experimental): Experimental milk protein based infant formula with varying carbohydrate and protein source
  Interventions: Other: milk protein formulas, varying carbohydrate/protein sources
- 4 (Experimental): Experimental milk protein based infant formula with varying carbohydrate and protein source
  Interventions: Other: milk protein formulas, varying carbohydrate/protein sources
- 5 (Experimental): Experimental milk protein based infant formula with varying carbohydrate and protein source
  Interventions: Other: milk protein formulas, varying carbohydrate/protein sources

INTERVENTIONS:
Other: milk protein formulas, varying carbohydrate/protein sources — ad lib for 0-8 days of age until 28 days of age

SUMMARY:
The objective of the study is to assess comparative gastrointestinal tolerance of normal term infants to various milk-protein infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infants; singleton birth; 37-42 weeks of age; >2490gms at birth; 0-8 days of age

Exclusion Criteria:

* medications/foods/formulas affecting GI tolerance;adverse medical history with possible effect on tolerance or growth

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 0-8 days of age until 28 days of age

SECONDARY OUTCOMES:
GI and intake parameters | 0-8 to 28 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Steven Davis, PhD, Study Director — Abbott Nutrition
Locations (15):
- United States (15):
  - Global Clinical Investigation, Aventura, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa, Coralville, Iowa
  - Medical Associates Clinic, Dubuque, Iowa
  - Kentucky Pediatric Research, Bardstown, Kentucky
  - PediaResearch, Inc, Owensboro, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Midwest Children's Health Research Institute, LLC, Lincoln, Nebraska
  - The Center for Human Nutrition, Omaha, Nebraska
  - MetroHealth Medical Center, Cleveland, Ohio
  - Pediatric Associates of Fairfield, Fairfield, Ohio
  - Ohio Pediatric Research Association, Huber Heights, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia